CLINICAL TRIAL: NCT04504045
Title: INFLAMMATION AND DRUG METABOLISM - Does the Effect of Drugs Decrease When Patients With Type 2 Diabetes Initiate Antidiabetic Treatment?
Brief Title: Metformin's Effect on Drug Metabolism in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment due to COVID-19, the study was stopped when recruited numbers fulfilled the pre-defined lower sample size.
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ann-Cathrine Dunvald, Principal Investigator, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AKF-395; 2020-000162-42 (EudraCT Number)
Record Dates: First submitted 2020-07-29; First posted 2020-08-07 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Caffeine; efavirenz; Losartan; Omeprazole; Metoprolol; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): Patients will receive metformin 1000-2000 mg daily for 12 weeks.
  Interventions: Drug: Metformin; Drug: Caffeine; Drug: Efavirenz; Drug: Losartan; Drug: Omeprazol; Drug: Metoprolol; Drug: Midazolam

INTERVENTIONS:
Drug: Metformin — 500 mg tablet
  Other Names: Glucose lowering treatment
Drug: Caffeine — As part of a 6-drug cocktail caffeine 100 mg tablet will be administered as a single dose before the initiation of metformin treatment and 3 weeks and 12 weeks after. The drug will be used as a probe to assess CYP1A2 activity.
Drug: Efavirenz — As part of a 6-drug cocktail efavirenz 50 mg coated tablet will be administered as a single dose before the initiation of metformin treatment and 3 weeks and 12 weeks after. The drug will be used as a probe to assess CYP2B6 activity.
Drug: Losartan — As part of a 6-drug cocktail losartan 12.5 mg coated tablet will be administered as a single dose before the initiation of metformin treatment and 3 weeks and 12 weeks after. The drug will be used as a probe to assess CYP2C9 activity.
Drug: Omeprazol — As part of a 6-drug cocktail Omeprazol 10 mg enteric-coated tablet will be administered as a single dose before the initiation of metformin treatment and 3 weeks and 12 weeks after. The drug will be used as a probe to assess CYP2C19 activity.
Drug: Metoprolol — As part of a 6-drug cocktail metoprolol 12.5 mg release tablet will be administered as a single dose before the initiation of metformin treatment and 3 weeks and 12 weeks after. The drug will be used as a probe to assess CYP2D6 activity.
Drug: Midazolam — As part of a 6-drug cocktail midazolam 2 mg oral solution will be administered as a single dose before the initiation of metformin treatment and 3 weeks and 12 weeks after. The drug will be used as a probe to assess CYP3A4 activity.

SUMMARY:
Type 2 diabetes is a major public health concern. It is widely established that type 2 diabetes in linked to activated innate immunity and increased levels of C-reactive protein and interleukin-6 (IL-6) in plasma. Studies in humans and in liver cells has shown that IL-6 downregulates important drug metabolizing enzymes in the liver (cytochrome P450 (CYP) enzymes). More than half of the most prescribed drugs are eliminated by biotransformation of these enzymes.

The investigators have previously shown that initiating glucose-lowering treatment (e.g. metformin, sulphonylureas and insulin) leads to decreased therapeutic efficacy of the blood-thinning vitamin-K antagonist warfarin. Due to the non-specific effect of glucose lowering drugs, the investigators hypothesize that this is caused by the glucose-lowering effect rather than drug-drug interactions caused by the individual drugs.

Based on the proposal that reversal of increased plasma glucose affects drug metabolism, the investigators will perform a clinical pharmacokinetic trial. The purpose of the study is to elucidate whether initiation of glucose-lowering treatment causes altered drug metabolism among patients with type 2 diabetes. The study will include newly diagnosed and untreated type 2 diabetes patients who will ingest a 6-drug cocktail consisting of probes for specific CYP enzymes. Plasma and urine will be drawn over 6 hours to determine concentrations of the drugs and their metabolites. Patients will then initiate metformin treatment and to assess both short- and long-term impact of glucose-lowering, the same 6-drug cocktail will be ingested, and concentrations measured, after three weeks and three months. To help understand the mechanism and the putative involvement of inflammation, markers of inflammation such as cytokines, transcription factors, etc. will also be assesses.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, not treated metformin.
* Hemoglobin 1Ac (HbA1c): ≥48 mmol/mol
* Age: 18-75 years
* Body Mass Index (BMI) ≤ 40 kg/m2
* Estimated Glomerular Filtration Rate (eGFR) > 60 mL/min
* Alanine Aminotransferase (ALAT), bilirubin and hemoglobin within reference range or clinically insignificant differ from this.

Exclusion Criteria:

* Acute or chronic infection or inflammation
* Active cancer
* Glutamic acid decarboxylase (GAD)-antibodies
* Known hypersensitivity to one or several of the drugs
* Intake of medications which can influence the safety of the patient or the results of the study
* Alcohol consumption above the limits recommended by the Danish Health Authorities (Men 14 units/week, women 7 units/week)
* Participation in other trials with interventions.
* Women: Positive pregnancy test at inclusion or on one of the test-days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Metabolic Rate of Midazolam (CYP3A4) at Week 3. | Baseline and Week 3.
  Change in activity of the drug metabolizing enzyme CYP3A4 following treatment with the glucose lowering drug metformin in 3 weeks. Assessment of the change is based on a change in the metabolic rate, which is the ratio between the concentration of midazolam and its primary metabolite is plasma (Probe drug for CYP3A4).
Change from Baseline in Metabolic Rate of Midazolam (CYP3A4) at Week 12. | Baseline and Week 12.
  Change in activity of the drug metabolizing enzyme CYP3A4 following treatment with the glucose lowering drug metformin in 12 weeks. Assessment of the change is based on a change in the metabolic rate, which is the ratio between the concentration of midazolam and its primary metabolite is plasma (Probe drug for CYP3A4).

SECONDARY OUTCOMES:
Change from Baseline in Metabolic Rate of Caffeine (CYP1A2) at Week 3. | Baseline and Week 3.
  Change in activity of the drug metabolizing enzymes CYP1A2 following treatment with the glucose lowering drug metformin after 3 weeks. The change in activity is based on the metabolic rate for the probe drug caffeine.
Change from Baseline in Metabolic Rate of Caffeine (CYP1A2) at Week 12. | Baseline and Week 12.
  Change in activity of the drug metabolizing enzymes CYP1A2 following treatment with the glucose lowering drug metformin after 12 weeks. The change in activity is based on the metabolic rate for the probe drug caffeine.
Change from Baseline in Metabolic Rate of Efavirenz (CYP2B6) at Week 3. | Baseline and Week 3.
  Change in activity of the drug metabolizing enzymes CYP2B6 following treatment with the glucose lowering drug metformin after 3 weeks. The change in activity is based on the metabolic rate for the probe drug Efavirenz.
Change from Baseline in Metabolic Rate of Efavirenz (CYP2B6) at Week 12. | Baseline and Week 12.
  Change in activity of the drug metabolizing enzymes CYP2B6 following treatment with the glucose lowering drug metformin after 12 weeks. The change in activity is based on the metabolic rate for the probe drug Efavirenz.
Change from Baseline in Metabolic Rate of Losartan (CYP2C9) at Week 3. | Baseline and Week 3.
  Change in activity of the drug metabolizing enzymes CYP2C9 following treatment with the glucose lowering drug metformin after 3 weeks. The change in activity is based on the metabolic rate for the probe drug Losartan.
Change from Baseline in Metabolic Rate of Losartan (CYP2C9) at Week 12. | Baseline and Week 12.
  Change in activity of the drug metabolizing enzymes CYP2C9 following treatment with the glucose lowering drug metformin after 12 weeks. The change in activity is based on the metabolic rate for the probe drug Losartan.
Change from Baseline in Metabolic Rate of Omeprazole (CYP2C19) at Week 3. | Baseline and Week 3.
  Change in activity of the drug metabolizing enzymes CYP2C19 following treatment with the glucose lowering drug metformin after 3 weeks. The change in activity is based on the metabolic rate for the probe drug Omeprazole.
Change from Baseline in Metabolic Rate of Omeprazole (CYP2C19) at Week 12. | Baseline and Week 12.
  Change in activity of the drug metabolizing enzymes CYP2C19 following treatment with the glucose lowering drug metformin after 12 weeks. The change in activity is based on the metabolic rate for the probe drug Omeprazole.
Change from Baseline in Metabolic Rate of Metoprolol (CYP2D6) at Week 3. | Baseline and Week 3.
  Change in activity of the drug metabolizing enzymes CYP2D6 following treatment with the glucose lowering drug metformin after 3 weeks. The change in activity is based on the metabolic rate for the probe drug Metoprolol.
Change from Baseline in Metabolic Rate of Metoprolol (CYP2D6) at Week 12. | Baseline and Week 12.
  Change in activity of the drug metabolizing enzymes CYP2D6 following treatment with the glucose lowering drug metformin after 12 weeks. The change in activity is based on the metabolic rate for the probe drug Metoprolol.
Change from Baseline in HbA1c at Week 3. | Baseline and Week 3.
  Change in the regulation of blood glucose over time assessed by HbA1c
Change from Baseline in HbA1c at Week 12. | Baseline and Week 12.
  Change in the regulation of blood glucose over time assessed by HbA1c
Change from Baseline in insulin resistance at Week 3. | Baseline and Week 3.
  An oral glucose tolerance test will be performed and glucose, insulin and c-peptide will be measured and combined by the Homeostatic Model Assessment (HOMA) to report insulin resistance.
Change from Baseline in insulin resistance at Week 12. | Baseline and Week 12.
  An oral glucose tolerance test will be performed and glucose, insulin and c-peptide will be measured and combined by the Homeostatic Model Assessment (HOMA) to report insulin resistance.
Change from Baseline in Interleukin-1-B at Week 3. | Baseline and Week 3.
  Change in patients inflammatory status assessed by measurement of Interleukin-1-B.
Change from Baseline in Interleukin-1-B at Week 12. | Baseline and Week 12.
  Change in patients inflammatory status assessed by measurement of Interleukin-1-B.
Change from Baseline in Interleukin-2 at Week 3. | Baseline and Week 3.
  Change in patients inflammatory status assessed by measurement of Interleukin-2.
Change from Baseline in Interleukin-2 at Week 12. | Baseline and Week 12.
  Change in patients inflammatory status assessed by measurement of Interleukin-2.
Change from Baseline in Interleukin-6 at Week 3. | Baseline and Week 3.
  Change in patients inflammatory status assessed by measurement of Interleukin-6.
Change from Baseline in Interleukin-6 at Week 12. | Baseline and Week 12.
  Change in patients inflammatory status assessed by measurement of Interleukin-6.
Change from Baseline in Interleukin-10 at Week 3. | Baseline and Week 3.
  Change in patients inflammatory status assessed by measurement of Interleukin-10.
Change from Baseline in Interleukin-10 at Week 12. | Baseline and Week 12.
  Change in patients inflammatory status assessed by measurement of Interleukin-10.
Change from Baseline in Interferon-a at Week 3. | Baseline and Week 3.
  Change in patients inflammatory status assessed by measurement of Interferon-a.
Change from Baseline in Interferon-a at Week 12. | Baseline and Week 12.
  Change in patients inflammatory status assessed by measurement of Interferon-a.
Change from Baseline in Interferon-B at Week 3. | Baseline and Week 3.
  Change in patients inflammatory status assessed by measurement of Interferon-B.
Change from Baseline in Interferon-B at Week 12. | Baseline and Week 12.
  Change in patients inflammatory status assessed by measurement of Interferon-B.
Change from Baseline in Interferon-y at Week 3. | Baseline and Week 3.
  Change in patients inflammatory status assessed by measurement of Interferon-y.
Change from Baseline in Interferon-y at Week 12. | Baseline and Week 12.
  Change in patients inflammatory status assessed by measurement of Interferon-y.
Change from Baseline in Tumor Necrosis Factor-a at Week 3. | Baseline and Week 3.
  Change in patients inflammatory status assessed by measurement of Tumor Necrosis Factor-a.
Change from Baseline in Tumor Necrosis Factor-a at Week 12. | Baseline and Week 12.
  Change in patients inflammatory status assessed by measurement of Tumor Necrosis Factor-a.
Change from Baseline in High Sensitivity C-Reactive Protein at Week 3. | Baseline and Week 3.
  Change in patients inflammatory status assessed by measurement of High Sensitivity C-Reactive Protein.
Change from Baseline in High Sensitivity C-Reactive Protein at Week 12. | Baseline and Week 12.
  Change in patients inflammatory status assessed by measurement of High Sensitivity C-Reactive Protein.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Cathrine Dunvald, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared due to general data protection regulation (GDPR).

REFERENCES:
- [Background] Stage TB, Pottegard A, Henriksen DP, Christensen MM, Hojlund K, Brosen K, Damkier P. Initiation of glucose-lowering treatment decreases international normalized ratio levels among users of vitamin K antagonists: a self-controlled register study. J Thromb Haemost. 2016 Jan;14(1):129-33. doi: 10.1111/jth.13187. Epub 2015 Dec 29. PMID 26559049
- [Derived] Dunvald AD, Nielsen F, Olsen DA, Ernst MT, Donnelly L, Soto-Pedre E, Kristiansen MR, Nielsen JS, Persson F, Hojlund K, Madsen JS, Sondergaard J, Pearson E, Pottegard A, Stage TB. Initiation of glucose-lowering drugs reduces the anticoagulant effect of warfarin-But not through altered drug metabolism in patients with type 2 diabetes. Br J Clin Pharmacol. 2023 Aug;89(8):2529-2541. doi: 10.1111/bcp.15725. Epub 2023 Apr 14. PMID 36967527